CLINICAL TRIAL: NCT06631391
Title: Pilot Study of Umbilical Cord Blood Natural Killer (NK) Cell Therapy for Pediatric Neuroblastoma.
Brief Title: Phase I Study of Umbilical Cord Blood Natural Killer (NK) Cell Therapy for Children With High-risk, R/R Neuroblastoma.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCBNK01
Record Dates: First submitted 2024-10-07; First posted 2024-10-08 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Neuroblastoma
Keywords: neuroblastoma, umbilical Cord blood NK cells
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Intervention Model Description: To evaluate the safety, tolerability and efficacy of umbilical cord blood natural killer cell injection in combination with other treatments (GD2 antibody, chemotherpay, etc) in high-risk, recurrent/refractory neuroblastoma in children
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with umbilical cord blood NK cells (Experimental): All subjects will receive Ex vivo Expanded and activated umbilical cord blood NK cells infusion.
  Interventions: Biological: umbilical cord blood NK cells

INTERVENTIONS:
Biological: umbilical cord blood NK cells — This is a phase I prospective clinical trial, including phase Ia and phase Ib. Phase Ia include 3 dose levels, utilizing a 3+3 design principle, and each dose level will enroll at least 3 subjects. The recommended dose for phase Ia was used in phase Ib. Each patient receives two courses of umbilical cord blood NK cell therapy (a total of 8 infusions of umbilical cord blood NK cells) and other therapy.

SUMMARY:
Neuroblastoma is the most common extracranial solid tumor, with more than half of the patients diagnosed at the metastatic stage, classified as high-risk. High-risk neuroblastoma has a poor prognosis and low survival rate. Despite treatment with induction, consolidation, and maintenance therapy including GD2 monoclonal antibody, the survival rate is only about 60%, and many patients still relapse, progress, and die.

NK cell therapy is an emerging immunotherapy that can effectively inhibit and kill tumor cells without significant adverse reactions, reducing the risk of tumor recurrence and metastasis, and improving patients' immunity and quality of life. Its safety has been widely recognized. Currently, clinical trials of NK cell infusion therapy for neuroblastoma patients are ongoing, and NK cell-based immunotherapy holds great clinical promise for neuroblastoma. We plan to conduct a phase I clinical trial on umbilical cord blood NK cell therapy in combination with other treatments (GD2 antibody, chemotherpay, etc) for high-risk, recurrent/refractory neuroblastoma in children to determine the maximum tolerated dose of umbilical cord blood NK cell therapy in these patients, thereby laying the foundation for future combination therapies and phase II and III clinical studies.

DETAILED DESCRIPTION:
To improve the prognosis of high-risk, Recurrent/Refractory neuroblastoma, we conducted a prospective Phase I clinical trial. Patients with high-risk and Recurrent/Refractory neuroblastoma who had undergone multidisciplinary treatment received umbilical cord blood NK cell infusions. The safety and efficacy of umbilical cord blood NK cells in combination with other therapy (GD2 antibody, chemotherpay, etc) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria must be met in order to be eligible for this trial:

1. Agree to participate in the trial and sign a written informed consent form;
2. Age ≤18 years, gender not limited;
3. Karnofsky (≥16 years old) or Lansky (<16 years old) physical status score (Appendix II) of at least 50;
4. Patients diagnosed with high-risk, recurrent/refractory neuroblastoma in children according to clinical diagnostic criteria, who have undergone comprehensive treatment (surgery, chemotherapy, radiotherapy ± stem cell transplantation ± GD2 monoclonal antibody therapy);
5. Expected survival period of at least 12 weeks;
6. The patient must have fully recovered from the acute toxic effects of all previous anticancer chemotherapy, such as recovery to grade I after bone marrow suppression;
7. Bone marrow suppressive chemotherapy: At least 21 days after the last bone marrow suppressive chemotherapy (if nitrosoureas were used previously, then 42 days);
8. Investigational drugs or anticancer therapies other than chemotherapy: Must not be used within 28 days before the planned start of NK cell immunotherapy. Full recovery from the clinically significant toxicity of that therapy must be confirmed;
9. Hematopoietic growth factors: At least 14 days after the last dose of long-acting growth factors or 3 days after the last dose of short-acting growth factors;
10. X-ray therapy (XRT): At least 14 days after local palliative XRT (small field port); if other substantial bone marrow (BM) irradiation is involved, including prior radioactive iodine metaiodobenzylguanidine (131I-MIBG) treatment, it must end at least 42 days ago;
11. Stem cell infusion without total body irradiation (TBI): No active graft-versus-host disease, must have ended at least 56 days after transplantation or stem cell infusion;
12. Laboratory tests during the screening period must meet the following conditions:

    1. Absolute neutrophil count (ANC) ≥1.0×10^9/L (if bone marrow involvement, then ANC ≥0.5×10^9/L)
    2. Platelet count (PLT) ≥75×10^9/L (if bone marrow involvement, then PLT ≥20×10^9/L)
    3. Bilirubin ≤1.5 times the upper limit of normal (ULN)
    4. Creatinine ≤1.5 times ULN (calculated using the standard Cockcroft-Gault formula)
    5. ALT/AST ≤3 times ULN (if there is liver metastasis, this can be relaxed to 5 times ULN)
13. During the study period, able to comply with outpatient treatment, laboratory monitoring, and necessary clinical visits; parents/guardians of pediatric or adolescent participants are capable of understanding, consenting to, and signing the informed consent form (ICF) and applicable child assent forms before initiating any protocol-related procedures; with parental/guardian consent, the participant is capable of expressing their consent (when applicable).

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for this trial:

1. Symptomatic brain metastases (patients whose brain metastases have been treated and whose symptoms have been stable for more than two months prior to enrollment may be enrolled, but must be confirmed by cranial MRI, CT, or venography as having no symptoms of cerebral hemorrhage);
2. Suffering from the following cardiovascular diseases: grade II or higher myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval ≥450 ms for males and ≥470 ms for females); according to the NYHA standard (Appendix Three), class III-IV heart failure, or echocardiography indicating left ventricular ejection fraction (LVEF) <50%;
3. Having a history of interstitial lung disease or suffering from interstitial lung disease at the same time;
4. Coagulation disorders (INR >1.5 or prothrombin time (PT) >ULN +4 seconds or APTT >1.5 ULN), with a tendency to bleed or currently receiving thrombolytic or anticoagulant therapy;
5. Arterial/venous thromboembolic events occurring within 12 months before enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
6. Known hereditary or acquired bleeding and thrombosis tendencies (such as hemophilia patients, coagulation disorders, thrombocytopenia, splenomegaly, etc.);
7. Long-term unhealed wounds or fractures (except pathological fractures caused by tumors);
8. Receiving major surgery or experiencing severe traumatic injuries, fractures, or ulcers within 4 weeks before enrollment;
9. Factors significantly affecting the absorption of oral medications, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
10. Experiencing abdominal fistula, gastrointestinal perforation, or abdominal abscess within 6 months before enrollment;
11. Routine urine tests showing proteinuria ≥ +, and confirmed 24-hour urine protein quantification ≥1.0 g;
12. Symptomatic serosal effusions requiring symptomatic treatment (including pleural effusion, ascites, pericardial effusion); Note: Asymptomatic serosal effusions can be enrolled, symptomatic serosal effusions after active symptomatic treatment (anticancer drugs cannot be used for treating serosal effusions), judged by the investigator to meet the enrollment criteria can be enrolled;
13. Active infections requiring antimicrobial treatment (e.g., needing antibacterial drugs, antiviral drugs, excluding chronic hepatitis B antiviral treatment, antifungal drug treatment);
14. History of psychoactive substance abuse that cannot be quit or has mental disorders;
15. Participated in other antitumor drug clinical trials within 4 weeks before enrollment;
16. Receiving systemic hormone therapy or undergoing any form of immunosuppressive therapy within 2 weeks before the first administration;
17. In the past 2 years, suffered from active autoimmune diseases requiring systemic treatment (such as using disease-modifying drugs, corticosteroids, or immunosuppressants); Note: Substitutive treatments (such as thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) do not count as systemic treatment;
18. Contraindications for IL-2 use;
19. Suffering from active infections requiring intravenous systemic treatment;
20. Vaccinated with live vaccines within one month before the first use of the study drug, seasonal influenza vaccination with inactivated virus vaccines is allowed, but intranasal attenuated live influenza vaccines are not allowed;
21. Previous or concomitant other uncured malignancies, cured skin basal cell carcinoma, cervical carcinoma in situ, and superficial bladder cancer are excluded;
22. Other conditions judged by the investigator that may affect the conduct of the clinical study and the determination of study results;
23. Virological tests during the screening period show any of the following:

    1. HBsAg positive and HBV DNA exceeds the upper limit of normal
    2. Anti-HCV positive and HCV RNA positive
    3. HIV positive
24. Undergone allogeneic tissue/organ transplantation;
25. Poor compliance, unable to cooperate with the clinical study.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of umbilical cord blood natural killer cell injection in combination with other treatments of high-risk, recurrent/refractory neuroblastoma in children | One weeks after the first cycle (each cycle is 28 days)
  According to the '3+3' design principle, the Maximum Tolerated Dose (MTD) is determined. Adverse events observed during the trial are graded according to the NCI CTCAE 5.0 criteria. Adverse events related to the drug (definitely related, probably related, or possibly related) occurring within 36 days after the first infusion of umbilical cord blood NK cells (during the first cycle) are considered as Dose-Limiting Toxicity (DLT). The definitions of DLT include:
  (1) Hematological toxicity:
  Grade 4 neutropenia lasting ≥7 days; Grade 4 thrombocytopenia lasting ≥7 days; (2) Grade 3/4 non-hematological toxicities (excluding nausea, vomiting, and alopecia); (3) Any toxicity leading to a delay in chemotherapy for more than 2 weeks.

SECONDARY OUTCOMES:
overall response rate (ORR) after 2 courses of umbilical cord blood natural killer cell infusion | Two weeks after the second cycle (a total of 16 weeks after the strart of first umbilical cord blood natural killer cell infusion)
  ORR was evaluated according to the International Neuroblastoma Response Criteria (INRC)

CONTACTS AND LOCATIONS:
Overall Officials: Yizhuo Zhang, Principal Investigator — SunYat Sen University Cancer Center
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou